CLINICAL TRIAL: NCT02771470
Title: Intestinal Microflora in Lung Cancer After Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2014SDU-QILU-G06
Record Dates: First submitted 2015-07-14; First posted 2016-05-13 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer; Effects of Chemotherapy; Tumor Immunity; Malnutrition
Keywords: Gut microflora; Lung cancer; Chemotherapy; Immunity; Nutrition
MeSH Terms: conditions — Lung Neoplasms; Malnutrition | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): Microbial composition using probiotics,3 capsules/times,3 times/day for 3 to 4 weeks
  Interventions: Drug: Probiotics
- Placebo (Placebo Comparator): Microbiota modulation using probiotics,3 capsules/times,3 times/day for 3 to 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Probiotics — Microbial composition using probiotic
  Other Names: containing clostridium butyricum
  Arms: Probiotic
Drug: placebo — Microbiota modulation using placebo
  Arms: Placebo

SUMMARY:
Probiotics modulate the gut microflora and immune status in lung cancer who need chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy destroys the intestinal mucosal barrier, affects intestinal flora, causing bacterial translocation, infection and other complications. Probiotics may restore the intestinal immunity, mucosal barrier and nutrient absorption.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for chemotherapy of lung cancer

Exclusion Criteria:

* Antibiotic, probiotic or prebiotic usage within 1month
* Other malignancy
* History of abdominal surgery
* Pregnant or breast-feeding (for females)
* Impaired liver or renal function
* Diabetes, thyroid disorder, coagulopathy or bleeding disorders, mental disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Composition of Microorganisms in stool after probiotic intervention | 2 months
  Primary coordination of fecal samples' 16s(%) rDNA will be compared between two groups using Braycurtis distance based Primary coordination analysis(PCoA)

SECONDARY OUTCOMES:
Frequency and severity of Adverse effects during Chemotherapy | 2 months
The change of immunity and nutrition index | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD.PhD., Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided